CLINICAL TRIAL: NCT05884528
Title: Assessment of Long-term Clinical Response to BoNT in Cervical Dystonia - Real-world Evidence of LongevitY of Botulinum Toxin in Cervical Dystonia
Brief Title: Assessment of Long-term Clinical Response to BoNT in Cervical Dystonia
Acronym: RELY-CD
Status: Completed | Type: Observational
Sponsor: Merz Therapeutics GmbH (Industry)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Organization: Merz Pharmaceuticals GmbH (Industry)
Other Study IDs: M602011073
Record Dates: First submitted 2023-05-08; First posted 2023-06-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cervical Dystonia
Keywords: spasmodic torticollis, focal dystonia
MeSH Terms: conditions — Torticollis; Dystonic Disorders | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; incobotulinumtoxinA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Complex-free BoNT/A formulation: Patients exclusively treated with the complex-free (CF) formulation (incobotulinumtoxinA). A maximum of 328 patients will be enrolled in this group.
  Interventions: Biological: CF BoNT/A
- Complex-containing BoNT/A formulations: Patients exclusively treated with a single complex-containing (CC) formulation (onabotulinumtoxinA or abobotulinumtoxinA). A maximum of 328 patients will be enrolled in this group.
  Interventions: Biological: CC BoNT/A
- Switcher CF to CC BoNT/A formulations: The CF to CC switcher group includes all patients that were switched from a CF to a CC BoNT/A formulation. If more than one switch occurred, the first switch determines the group. Both switcher groups will in sum not exceed 325 patients.
  Interventions: Biological: CF to CC BoNT/A
- Switcher CC to CF BoNT/A formulations: The CC to CF switcher group includes all patients that were switched from a CC to a CF BoNT/A formulation. If more than one switch occurred, the first switch determines the group. Both switcher groups will in sum not exceed 325 patients.
  Interventions: Biological: CC to CF BoNT/A

INTERVENTIONS:
Biological: CC BoNT/A — Complex-containing BotulinumtoxinA (BoNT/A) formulations
  Other Names: onabotulinumtoxinA; abobotulinumtoxinA
  Groups: Complex-containing BoNT/A formulations
Biological: CF BoNT/A — Complex-free BotulinumtoxinA (BoNT/A) formulation
  Other Names: incobotulinumtoxinA; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Groups: Complex-free BoNT/A formulation
Biological: CF to CC BoNT/A — Switch from complex-free to complex-containing BoNT/A formulations
  Other Names: incobotulinumtoxinA; onabotulinumtoxinA; abobotulinumtoxinA
  Groups: Switcher CF to CC BoNT/A formulations
Biological: CC to CF BoNT/A — Switch from complex-containing to complex-free BoNT/A formulations
  Other Names: onabotulinumtoxinA; abobotulinumtoxinA; incobotulinumtoxinA
  Groups: Switcher CC to CF BoNT/A formulations

SUMMARY:
The goal of this retrospective, international, multi-center chart abstraction is to learn about the long-term impact of product-specific immunogenicity-related factors in different botulinum neurotoxin type A formulations in patients suffering from cervical dystonia. The main question it aims to answer is:

Do complex-containing (CC) botulinum toxin formulations impact the long-term clinical outcome in cervical dystonia patients compared to a complex-free (CF) formulation?

Researchers will compare differences observed in years 2 and 7 between two toxin groups, i.e., botulinum neurotoxins type A containing complexing proteins (CC) and without complexing proteins (CF).

DETAILED DESCRIPTION:
Botulinum neurotoxin type A (BoNT/A) is first-line treatment in patients suffering from cervical dystonia. Effect of BoNT/A is temporary and must be repeated to maintain clinical effect. As for all biologics, repeated treatment bears the risk of activating an immune response due to the immunogenic nature of foreign proteins. Clinical signs of a potential immune response are reduced, or loss of efficacy, decreased duration of effect, and the need of a dose increase to maintain effect. Due to the different degree of purity and protein content, it is reasonable to assume that commercial BoNT/A formulations differ in immunogenic properties.

Pivotal clinical trials and monocentric real-world studies demonstrated an increased incidence of neutralizing antibodies (NAbs) and NAb-associated partial or complete secondary non-response. However, the clinical relevance of potential immunogenicity-related mechanisms has not been demonstrated in a larger multicentric cohort in a real-world setting. This chart abstraction is designed to address this gap.

ELIGIBILITY:
* Clinical diagnosis of cervical dystonia
* Adults (m/f) 18-64 years of age at start of BoNT/A treatment
* Patient's written informed consent if required by local and/or national law.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will comprise of patients with a diagnosis of cervical dystonia who received regular BoNT/A injections for symptomatic treatment of the disease. The sub-populations consist of long-term patients treated with only ever one BoNT/A formulation (monotherapy) or 2 BoNT/A formulations (switcher).
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2023-07-08 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a clinically meaningful change in dose-effect at year 7 compared to reference year 2 between complex-free and complex-containing BoNT/A monotherapy | Year 2 and year 7
  Dose-effect is a change in treatment response following dose adjustment.

SECONDARY OUTCOMES:
Clinical meaningfulness of change in efficacy from baseline (first visit on record) at each visit in years 2, 5, 7, 10 in all treatment groups | Baseline (first visit on record), years 2, 5, 7, and 10

OTHER OUTCOMES:
Incidence of frequent AEs overall and in patients with altered dose-effect | Years 2, 5,7, and 10
Health-related quality of life measured by the EQ-5D | Years 2, 5,7, and 10
Health-related quality of life measured by the SF-36 | Years 2, 5,7, and 10
Health-related quality of life measured by the CDQ24 | Years 2, 5,7, and 10
Sub-analysis of all outcome measures in switcher population (patients treated with more than one BoNT/A formulation) | Years 2, 5,7, and 10

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Therapeutics
Locations (1):
- Düsseldorf University Hospital, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware JE Jr, Kosinski M, Gandek B, Aaronson NK, Apolone G, Bech P, Brazier J, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. The factor structure of the SF-36 Health Survey in 10 countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1159-65. doi: 10.1016/s0895-4356(98)00107-3. PMID 9817133
- [Background] Albanese A, Bhatia K, Bressman SB, Delong MR, Fahn S, Fung VS, Hallett M, Jankovic J, Jinnah HA, Klein C, Lang AE, Mink JW, Teller JK. Phenomenology and classification of dystonia: a consensus update. Mov Disord. 2013 Jun 15;28(7):863-73. doi: 10.1002/mds.25475. Epub 2013 May 6. PMID 23649720
- [Background] Albrecht P, Jansen A, Lee JI, Moll M, Ringelstein M, Rosenthal D, Bigalke H, Aktas O, Hartung HP, Hefter H. High prevalence of neutralizing antibodies after long-term botulinum neurotoxin therapy. Neurology. 2019 Jan 1;92(1):e48-e54. doi: 10.1212/WNL.0000000000006688. Epub 2018 Nov 21. PMID 30464031
- [Background] Carr WW, Jain N, Sublett JW. Immunogenicity of Botulinum Toxin Formulations: Potential Therapeutic Implications. Adv Ther. 2021 Oct;38(10):5046-5064. doi: 10.1007/s12325-021-01882-9. Epub 2021 Sep 13. PMID 34515975